CLINICAL TRIAL: NCT05300217
Title: Evaluating the Efficacy and the Acceptability of the Website "Ich Bin Alles" to Improve Depression Literacy in Adolescents
Brief Title: Evaluation of a Website to Improve Depression Literacy in Adoldescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20115_2
Record Dates: First submitted 2022-03-10; First posted 2022-03-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder; Depression in Adolescence
Keywords: Knowledge; Mental Health; Depression Literacy; Website; Online; Adolescence; Youth
MeSH Terms: conditions — Depressive Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two intervention groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants are not aware of the assigned intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group 1 - Strategies for promoting mental health (Experimental): Exposure to information about strategies for promoting mental health
  Interventions: Other: Strategies for promoting mental health
- Intervention Group 2 - General information about depression (Experimental): Exposure to general information about depression
  Interventions: Other: General information about depression

INTERVENTIONS:
Other: Strategies for promoting mental health — Before starting the intervention, the participants are told that they will be shown parts of a website about depression. The participants are instructed to carefully attend to the website (e.g., to read the text precisely, to hear attentively to the podcasts and images on the website). The time window spent for the reception of each part of the website are fixed.
  The participants in this intervention group will only be shown parts of the website regarding strategies for promoting mental health
  Arms: Intervention Group 1 - Strategies for promoting mental health
Other: General information about depression — Before starting the intervention, the participants are told that they will be shown parts of a website about depression. The participants are instructed to carefully attend to the website (e.g., to read the text precisely, to hear attentively to the podcasts and to view carefully the videos and images on the website). The time window spent for the reception of each part of the website are fixed.
  The participants in this intervention group will only be shown parts of the website regarding general information about depression
  Arms: Intervention Group 2 - General information about depression

SUMMARY:
The aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy (knowledge about depression, which aid the recognition, treatment or prevention of depression) in healthy adolescents. The investigators will examine whether the website improves depression literacy in healthy adolescents aged 12 to 18 years. The investigators will also assess the acceptability of the website among adolescents.

DETAILED DESCRIPTION:
Few young people with major depressive disorder seek professional treatment in time. Concerns about social stigma, confidentiality, and limited knowledge about mental health conditions, such as depression, or mental health services are some of the main barriers to seek treatment. To address these problems, we developed an evidence-based website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy.

To improve depression literacy, the website provides general information about depression as psychiatric disorder in adolescents (e.g., symptoms, causes, course and treatment of depression). Furthermore, the website provides information about self-help strategies for depression and prevention of depression; i.e., strategies for promoting mental health (e.g., reducing stress, doing exercise, undertaking positive activities), which are meant to serve as an addition to professional treatments of depression or to promote mental health in adolescents.

Target groups of the website are adolescents aged 12 to 18 years seeking help for depression, as well as healthy adolescents seeking information about mental health promotion or depression. Easy access to information about depression would make early recognition of depression more likely and engage young people to seek help for depression.

Since the website targets two different groups, the investigators will evaluate the website accordingly:

Target group 1: Adolescents with a major depressive disorder (acute or remitted) Target group 2: Healthy Adolescents (no mental health condition) The current study will focus on target group 2. A study focusing on target group 1 can be found in a separately registered clinical trial on clinicaltrials.gov.

The primary aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy in healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

- Intelligence quotient (IQ) of ≥ 80

Exclusion Criteria:

* Current diagnosis of a mental disorder
* Remitted depressive disorder
* Insufficient knowledge of German

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Depression Literacy - Strategies for promoting mental health | Pre-Test, Post-Test (within 2 hours), Follow-Up 1 (Week 2), Follow-Up 2 (Week 4)
  This self-designed questionnaire is a self-report inventory to assess knowledge of strategies for promoting mental health (exercise, dealing with problems and stress, positive attitude, postive activities and social contacts; 27 items), with higher scores indicating more knowledge of strategies for promoting mental health. Participants will complete this self-designed questionnaire at pre-test, post-test and the two follow-ups to determine change in knowledge of strategies for promoting mental health.
Depression Literacy - Depression as psychiatric disorder | Pre-Test, Post-Test (within 2 hours), Follow-Up 1 (Week 2), Follow-Up 2 (Week 4)
  This self-designed questionnaire is a self-report inventory to assess knowledge of depression as psychiatric disorder (frequency and comorbidities, treatment, symptoms, causes and course of depression; 27 items), with higher scores indicating more knowledge of depression as psychiatric disorder. Participants will complete this self-designed questionnaire at pre-test, post-test and the two follow-ups to determine change in knowledge of depression as psychiatric disorder

SECONDARY OUTCOMES:
Visual Aesthetics of Websites Inventory Short Version (VisAWI-S) | Post-Test (within 2 hours)
  The short version of the Visual Aesthetics of Websites Inventory (VisAWI-S) is self-report inventory to assess the evaluation of the website's design - especially the perceived visual aesthetics. Participants indicated their response to the four items (e.g., "The layout appears professionally designed") on a seven-point Likert scale (ranging from 1 "do not agree at all" to 7 "do fully agree")
Overall reception of the website | Post-Test (within 2 hours)
  The overall reception of the website as measured with a self-designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Professor, Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive patient information, such as sociodemographic information and comorbidities. Since patients could possibly be identified by making our raw data publicly available, ethical principles of protecting patient confidentiality would be breached. Aggregated group data can be made available upon request.

REFERENCES:
- [Derived] Kloek MWH, Zsigo C, Primbs R, Iglhaut L, Kaubisch S, Piechaczek CE, Keim PM, Feldmann L, Schulte-Korne G, Greimel E. Improving adolescents' knowledge about mental health and depression: a randomized experimental study of web-based information. Front Digit Health. 2025 Nov 18;7:1640366. doi: 10.3389/fdgth.2025.1640366. eCollection 2025. PMID 41341464